CLINICAL TRIAL: NCT06418711
Title: ICoN-1: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Efficacy and Safety of Clofazimine Inhalation Suspension When Added to Guideline-Based Therapy in Participants With Nontuberculous Mycobacterial Infection
Brief Title: ICoN-1 Phase 3 Study of the Efficacy and Safety of Treatment With MNKD-101, Clofazimine Inhalation Suspension
Acronym: ICoN-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKC-CI-002
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: MAC Lung Disease; Treatment Refractory MAC Lung Disease; Mycobacterium Infections, Nontuberculous
Keywords: Bronchiectasis; NTM (Nontuberculous mycobacteria); MAC (Mycobacterium avium complex); MABSC (Mycobacterium abscessus complex); Pulmonary Nontuberculous Mycobacteria; Respiratory Infection; antimycobacterial activity; antimycobacterial therapy; MAC infections; MAC Lung disease; MAC pulmonary infection; Mycobacteria; mycobacterium; Mycobacterium Avium Complex Infections; Mycobacterium avium complex lung disease; mycobacterium Infections; Nontuberculous; Non-tuberculous mycobacterial (NTM) infections; Nontuberculous mycobacterial lung disease; Non-tuberculous mycobacterial pulmonary disease; NTM infection; NTM lung disease; NTM Pulmonary Disease; NTM lung infection; Pulmonary MAC disease; Pulmonary Mycobacterium Avium Complex disease; Treatment refractory MAC lung disease; Treatment refractory mycobacterial lung disease; Treatment refractory NTM lung infection; Treatment refractory NTM pulmonary disease; Respiratory Tract diseases; Actinomycetales Infections; Gram-Positive Bacterial Infections; Bacterial Infections; Bacterial Infections and Mycoses; Infections; Mycobacterium Infections, Nontuberculous; Mycobacterium avium-intracellulare Infection; Lung diseases; Anti-Bacterial Agents; Anti-infective Agents; Antitubercular Agents; Azithromycin; Amikacin; Ethambutol; Clofazimine; Lamprene
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous; Bronchiectasis; Mycobacterium avium-intracellulare Infection; Respiratory Tract Infections; Mycobacterium Infections; Infections; Respiratory Tract Diseases; Actinomycetales Infections; Gram-Positive Bacterial Infections; Bacterial Infections; Bacterial Infections and Mycoses; Lung Diseases

STUDY DESIGN:
Intervention Model Description: At least 234 eligible participants will be randomized in a 2:1 ratio of 1 of 2 possible treatment assignments in order to ensure that a minimum of 180 participants are evaluable for efficacy: Clofazimine Inhalation Suspension (N=120) and placebo (n=60). Randomization will be stratified by type of nontuberculous mycobacteria (NTM) infection (Mycobacterium avium complex [MAC] infection only vs MAC co-infection with Mycobacterium abscessus complex [MABSC] or other NTM species) based on historical samples used to establish eligibility during screening. Enrollment of participants with MAC coinfection with MABSC or other NTM species will be capped at 20% of all participants to limit heterogeneity in the participant population.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During Part A of the study, the identity of the treatments will be concealed by the use of a placebo, and treatment unblinding will only occur in the case of participant emergencies or if requested by the Data and Safety Monitoring Board (DSMB).
  Sputum Test Results: Results of post-baseline testing for the presence of NTM in sputum will remain concealed until the participant has completed Part A of the study and the participant's result for the sample taken at the end of Month 6 becomes available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clofazimine Inhalation Suspension (Experimental): MNKD-101 (Clofazimine Inhalation Suspension) is a micronized suspension with a concentration of 20 mg/mL. Study drug will be inhaled using the PARI breath-enhanced jet nebulizer system daily for 28 days in Cycle 1. Cycle 2 will commence after 56 days off treatment and resume daily for 28 days. Dose: 80 mg
  Interventions: Drug: Clofazimine Inhalation Suspension
- Placebo (Placebo Comparator): The placebo is comprised of isotonic saline (0.9% weight/volume sodium chloride). Study drug will be inhaled using the PARI breath-enhanced jet nebulizer system daily for 28 days in Cycle 1. Cycle 2 will commence after 56 days off treatment and resume daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clofazimine Inhalation Suspension — Eligible participants will be randomized in a 2:1 ratio to 1 of 2 possible treatment assignments, Clofazimine Inhalation Suspension or Placebo.
  Other Names: MNKD-101
  Arms: Clofazimine Inhalation Suspension
Drug: Placebo — Eligible participants will be randomized in a 2:1 ratio to 1 of 2 possible treatment assignments, Clofazimine Inhalation Suspension or Placebo.
  Arms: Placebo

SUMMARY:
This clinical trial is designed to compare the efficacy and safety of Clofazimine Inhalation Suspension versus placebo when added to guideline-based therapy (GBT)

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study (Part A) designed to compare the efficacy and safety of Clofazimine Inhalation Suspension versus placebo when added to guideline-based therapy (GBT). The primary objective of this study will be to compare the efficacy of Clofazimine Inhalation Suspension versus placebo as assessed by the co-primary endpoints, sputum culture conversion and change in Quality of Life-Bronchiectasis Respiratory Symptoms Score (QoL-B RSS).

An open label extension study (Part B) will be offered to qualified participants for treatment with Clofazimine Inhalation Suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of signed and dated informed consent document(s) indicating the participant has been informed of all pertinent aspects of the trial.
2. Age ≥18 years or legal age for the participating country (e.g., the legal age in South Korea is 19 years) and ≤85 years.
3. Evidence of underlying nodular bronchiectasis and/or fibrocavitary disease on a chest radiograph or chest computed tomography, as determined by the investigator, within the last 12 months.
4. MAC-positive culture results from at least two separates (at least 1 week apart) expectorated sputum samples, one taken within 12 months, and another taken within 3 months prior to the date of informed consent. Note: A sputum culture will be obtained at baseline, but the participant may be randomized prior to availability of the results.
5. Be able to produce at least 3 mL of sputum or be willing to undergo an induction that produces at least 3 mL of sputum for mycobacteriology.
6. FEV1 ≥40% of predicted during screening, as calculated by the local spirometry laboratory standards.
7. Currently receiving a multi-drug regimen of GBT for pulmonary NTM infection in line with the 2020 ATS/ERS/ESCMID/IDSA guideline for the treatment of NTM pulmonary disease for at least 6 months prior to consenting in this study, with no changes in this regimen within 2 months of screening.
8. For female participants of childbearing potential, a negative serum pregnancy test and agreement to use a protocol-recommended method of contraception during heterosexual intercourse from the start of the screening period until ≥12 months after the final dose of study therapy. Note: A female participant is considered to be of childbearing potential, i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
9. For male participants who can father a child and are having intercourse with females of childbearing potential, agreement to use a protocol-recommended method of contraception from the start of the study therapy until ≥12 months after the final dose of study therapy and to refrain from sperm donation from the start of study therapy until ≥12 months after administration of the final dose of study therapy. Note: A male participant is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.
10. Willingness and ability to comply with scheduled visits, drug inhalation plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

1. Cystic fibrosis.
2. Active tuberculosis. Note: Participants with a history of treated latent or active tuberculosis may be eligible as long as their sputum cultures in the last year are negative for tuberculosis and they are deemed by the investigator as not having current active tuberculosis.
3. Disseminated MAC or MABSC infection or participants with isolated MABSC infection.
4. Recent (i.e., within the last 3 months from date of screening) ICU admission with or without mechanical ventilation.
5. Inability to inhale with a nebulizer, in the opinion of the investigator.
6. Participants with known hypersensitivity to any of the ingredients or excipients of clofazimine.
7. Prior therapy with clofazimine in the previous 4 months from date of screening.
8. Participants with known resistance to clofazimine as treatment for MAC (i.e., MIC >8 ug/mL for MAC).
9. Prior therapy with amikacin by any route of administration (e.g., inhaled or IV) in the previous 2 months from date of screening.
10. Ongoing participation in any other interventional drug or device clinical trial, or exposure to another investigational drug within 28 days prior to start of study treatment. Note: For investigational therapies that have a prolonged half-life, a case-by-case assessment will be made regarding the required washout period prior to being eligible for this study.
11. Current (or planned during the study) pregnancy or breastfeeding.
12. QT prolongation during screening (450 ms or longer), and/or uncontrolled sinus rhythm (>110/minute).
13. Increased risk of proarrhythmia (e.g., recent [within 6 months] myocardial infarction, stroke, heart failure decompensation or left ventricular ejection of <45%, ventricular arrhythmias, torsade de pointes, unstable angina, or high-degree atrioventricular block).
14. A family history of sudden cardiac death, unexplained death, long-QT syndrome, or death from a primary dysrhythmia potentially associated with QT prolongation.
15. Recent (within 6 months) initiation of or change in the dosing regimen of any concomitant medication that is known to prolong the QT interval. Note: Participants who are on a stable regimen, in the opinion of the investigator, of the concomitant medication during screening are eligible.
16. Chronic and clinically meaningful, in the opinion of the investigator, abnormalities in potassium, magnesium, or calcium levels.
17. Active pulmonary malignancy (primary or metastatic) or any malignancy requiring chemotherapy or radiation therapy within 3 years before screening or anticipated during the study period.
18. Current alcohol, medication, or illicit drug abuse.
19. Prior or ongoing social or medical condition (e.g., concomitant illness, psychiatric condition, behavioral disorder), medical history, physical findings, ECG findings or laboratory abnormality that, in the opinion of the investigator, could adversely affect the safety of the participant, makes it unlikely that the course treatment or follow-up would be completed, or could impair the assessment of study results.
20. Any prior use of bedaquiline within 1 year of screening.
21. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN) or total bilirubin >1.5 times ULN during screening.
22. Absolute neutrophil count <500/µL during screening.
23. Use of prednisone ≥10mg/day within 3 months prior to screening, or other significant immunosuppression as deemed by the investigator.
24. Estimated glomerular filtration rate <30mL/minute/1.73 m2 (according to the CKD-EPI 2021 creatine equation) during screening.
25. Advanced liver disease (Child-Pugh Class A, B, or C).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
(Part A) Sputum culture conversion (i.e., 3 consecutive monthly sputum cultures negative for MAC) by the end of Month 6 | Baseline to the end of Month 6
  (Part A) Sputum culture conversion (i.e., 3 consecutive monthly sputum cultures negative for MAC) by the end of Month 6 (Part A)
(Part A) Change in QoL-B RSS from baseline to end of Month 6 (Part A) | Baseline to end of Month 6
  (Part A) Change in QoL-B RSS from baseline to end of Month 6 (Part A)

SECONDARY OUTCOMES:
(Part A) Time to a composite endpoint of pulmonary worsening, as defined by: all-cause mortality, respiratory-related hospitalization, or the requirement for parenteral (inhaled or IV) antibiotic use for NTM or other pneumonia treatment (Part A) | Baseline to the end of Month 6
  (Part A) Time to a composite endpoint of pulmonary worsening, defined as the occurrence of any of the following clinical events: all-cause mortality, respiratory-related (as determined by the investigator) hospitalization, or the requirement for parenteral (inhaled or IV) antibiotic use for NTM or other pneumonia treatment (Part A)
(Part A) Change in 6-minute walk distance (6MWD) from baseline to the end of Month 6 | Baseline to the end of Month 6
  (Part A) Change in 6-minute walk distance (6MWD) from baseline to the end of Month 6
(Part A) Change in participant identified Most Bothersome Symptom (MBS) from baseline to the end of Month 6 | Baseline to the end of Month 6
  (Part A) Change in participant identified Most Bothersome Symptom (MBS) from baseline to the end of Month 6
(Part A) Change in response to the Patient Global Impression of Severity (PGI-S) questionnaire from baseline to the end of Month 6 | Baseline to the end of Month 6
  (Part A) Change in response to the Patient Global Impression of Severity (PGI-S) questionnaire from baseline to the end of Month 6
(Part A) Response to the Patient Global Impression of Change (PGI-C) questionnaire at the end of Month 6 | Baseline to the end of Month 6
  (Part A) Response to the Patient Global Impression of Change (PGI-C) questionnaire at the end of Month 6

OTHER OUTCOMES:
(Part A) Sputum MAC density in CFU/mL at the end of Month 6 | End of Month 6
  (Part A) Sputum MAC density in CFU/mL at the end of Month 6
(Part A) Sputum MAC resistance patterns at the end of Month 6, measured using sputum microbiological lab assessments | End of Month 6
  (Part A) Sputum MAC resistance patterns at the end of Month 6, measured using sputum microbiological lab assessments
(Part A) Time to first negative MAC sputum culture in participants who achieve culture conversion by Month 6 | End of Month 6
  (Part A) Time to first negative MAC sputum culture in participants who achieve culture conversion by Month 6
(Part A) Time to sputum culture conversion in participants who achieve culture conversion by Month 6 | End of Month 6
  (Part A) Time to sputum culture conversion in participants who achieve culture conversion by Month 6
(Part A) Rate of sputum culture conversion (MAC-negative to MAC-positive) in the subgroup of study participants whose baseline sputum culture is negative for NTM | Baseline to end of study
  (Part A) Rate of sputum culture conversion (MAC-negative to MAC-positive) in the subgroup of study participants whose baseline sputum culture is negative for NTM
(Part A) Time-to-positivity (TTP) in broth cultures for MAC in sputum at the end of Months 1,2,3,4,5, and 6 | End of Months 1,2,3,4,5, and 6
  (Part A) Time-to-positivity (TTP) in broth cultures for MAC in sputum at the end of Months 1,2,3,4,5, and 6
(Part A) Changes in inflammatory markers (specific tests to be determined) from baseline to the end of Months 1,3,4, and 6 | End of Months Months 1,3,4, and 6
  (Part A) Changes in inflammatory markers (specific tests to be determined) from baseline to the end of Months 1,3,4, and 6
(Part A) Rate of pulmonary worsening, as diagnosed and defined by the investigator based upon a participant's need for a limited course of antibiotic medication to treat an acute worsening of symptoms, in Months 1,2,3,4,5, and 6 | End of Months 1,2,3,4,5, and 6
  (Part A) Rate of pulmonary worsening, as diagnosed and defined by the investigator based upon a participant's need for a limited course of antibiotic medication to treat an acute worsening of symptoms, in Months 1,2,3,4,5, and 6
(Part A) Rate of respiratory-related (as defined by the investigator) hospitalization | Baseline to end of Month 6
  (Part A) Rate of respiratory-related (as defined by the investigator) hospitalization
(Part A) All-cause mortality | Baseline to end of Month 6
  (Part A) All-cause mortality
(Part A) Respiratory-related (as determined by the investigator) mortality | Baseline to end of Month 6
  (Part A) Respiratory-related (as determined by the investigator) mortality
(Part A) Use of rescue medication (i.e., initiation of anti-mycobacterial medication that is recommended by the investigator due to a perception of lack of efficacy of study drug) for pulmonary NTM infection | Baseline to end of Month 6
  (Part A) Use of rescue medication (i.e., initiation of anti-mycobacterial medication that is recommended by the investigator due to a perception of lack of efficacy of study drug) for pulmonary NTM infection
(Part A) Difference in days of absenteeism from work | Baseline to end of Month 6
  (Part A) Difference in days of absenteeism from work
(Part A) Difference in hospitalization days | Baseline to end of Month 6
  (Part A) Difference in hospitalization days
(Part A) Difference in number of emergency room visits | Baseline to end of Month 6
  (Part A) Difference in number of emergency room visits
(Part A) Difference in number of urgent care visits | Baseline to end of Month 6
  (Part A) Difference in number of urgent care visits
(Part A) Difference in number of unscheduled doctor visits | Baseline to end of Month 6
  (Part A) Difference in number of unscheduled doctor visits
(Part A) Change in BMI from baseline to the end of Month 6 | Baseline to end of Month 6
  (Part A) Change in BMI from baseline to the end of Month 6
(Part A) Slope of the change from baseline to end of Month 6 in log10 CFU/mL of MAC | Baseline to end of Month 6
  (Part A) Slope of the change from baseline to end of Month 6 in log10 CFU/mL of MAC
(Part A) Changes in other QoL-B questionnaire domain (Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden) scores from baseline to the end of Month 6 | Baseline to the end of Month 6
  (Part A) Changes in other QoL-B questionnaire domain (Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden) scores from baseline to the end of Month 6
(Part A) Changes in shortness of breath when sitting or at rest and when exercising from baseline to the end of Month 6, measured using stand-alone shortness of breath questionnaire | Baseline to the end of Month 6
  (Part A) Changes in shortness of breath when sitting or at rest and when exercising from baseline to the end of Month 6, measured using stand-alone shortness of breath questionnaire
(Part A) Change in most severe symptom at baseline from baseline to the end of Month 6, measured using stand-alone shortness of breath questionnaire | Baseline to the end of Month 6
  (Part A) Change in most severe symptom at baseline from baseline to the end of Month 6, measured using stand-alone shortness of breath questionnaire
(Part A) Concentration of clofazimine in plasma | Baseline to end of Month 6
  (Part A) Concentration of clofazimine in plasma
(Part A) Change in forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) from baseline to the end of Month 6 | Baseline to the end of Month 6
  (Part A) Change in forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) from baseline to the end of Month 6
(Part A) Rate of study drug discontinuations | Baseline to end of Month 6
  (Part A) Rate of study drug discontinuations
(Part A) Rate of study drug dose reductions | Baseline to end of Month 6
  (Part A) Rate of study drug dose reductions
(Part A) Rate of treatment-emergent adverse events (TEAEs) | Baseline to end of Month 6
  (Part A) Rate of treatment-emergent adverse events (TEAEs)
(Part A) Rate of treatment-related adverse events (TRAEs) | Baseline to end of Month 6
  (Part A) Rate of treatment-related adverse events (TRAEs)
(Part A) Rate of serious adverse events (SAEs) | Baseline to end of Month 6
  (Part A) Rate of serious adverse events (SAEs)
(Part A) Rate of laboratory abnormalities | Baseline to end of Month 6
  (Part A) Rate of laboratory abnormalities
(Part A) Rate of electrocardiogram (ECG) abnormalities | Baseline to end of Month 6
  (Part A) Rate of electrocardiogram (ECG) abnormalities
(Part B) Adverse Events (AEs) related to inhalation intolerability | Study Month 7 through Study Month 22
  (Part B) Adverse Events (AEs) related to inhalation intolerability
(Part B) AEs due to skin discoloration | Study Month 7 through Study Month 22
  (Part B) AEs due to skin discoloration
(Part B) AEs due to QTc changes | Study Month 7 through Study Month 22
  (Part B) AEs due to QTc changes
(Part B) Sputum culture conversion (i.e., 3 consecutive- monthly sputum cultures negative for NTM | Study Month 7 through Study Month 22
  (Part B) Sputum culture conversion (i.e., 3 consecutive- monthly sputum cultures negative for NTM
(Part B) Rate of sputum culture conversion (MAC-negative to MAC-positive) in the subgroup of study participants whose baseline sputum culture is negative | Study Month 7 through Study Month 22
  (Part B) Rate of sputum culture conversion (MAC-negative to MAC-positive) in the subgroup of study participants whose baseline sputum culture is negative
(Part B) Rate of persistency of negative sputum culture | Study Month 7 through Study Month 22
  (Part B) Rate of persistency of negative sputum culture
(Part B) Change in QoL-B RSS from baseline | Study Month 7 through Study Month 22
  (Part B) Change in QoL-B RSS from baseline
(Part B) Difference in days of absenteeism from work | Study Month 7 through Study Month 22
  (Part B) Difference in days of absenteeism from work
(Part B) Difference in hospitalization days | Study Month 7 through Study Month 22
  (Part B) Difference in hospitalization days
(Part B) Difference in number of emergency room visits | Study Month 7 through Study Month 22
  (Part B) Difference in number of emergency room visits
(Part B) Difference in number of urgent care visits | Study Month 7 through Study Month 22
  (Part B) Difference in number of urgent care visits
(Part B) Difference in number of unscheduled doctor visits | Study Month 7 through Study Month 22
  (Part B) Difference in number of unscheduled doctor visits
(Part B) Sustainability of response to Clofazimine Inhalation Suspension, evaluated quarterly while on treatment following initial conversion, for participants who convert | Study Month 7 through Study Month 22
  (Part B) Sustainability of response to Clofazimine Inhalation Suspension, evaluated quarterly while on treatment following initial conversion, for participants who convert. Culture conversion with sustainability is defined as achieving culture conversion and then having no more than 2 consecutive broth or Agar positive sputum cultures and no Agar positive culture observed once initial conversion is achieved.
(Part B) Durability of response to Clofazimine Inhalation Suspension, evaluated quarterly following active treatment, for participants who remain converters at the end of active treatment | Study Month 7 through Study Month 22
  (Part B) Durability of response to Clofazimine Inhalation Suspension, evaluated quarterly following active treatment, for participants who remain converters at the end of active treatment. Culture conversion with durability is defined as achieving culture conversion and remaining a converter at the end of active treatment and then having no broth or Agar positive sputum culture following active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Fares, MD, Study Director — Mannkind Corporation
Locations (99):
- United States (54):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - University of California San Francisco Fresno, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Hospital, Newport Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford University, Stanford, California
  - National Jewish Health, Denver, Colorado
  - UCONN Health, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - VA Bay Pines, Bay Pines, Florida
  - St. Francis Sleep, Allergy & Lung Institute, Clearwater, Florida
  - Malcolm Randall Veterans Affairs Medical Center, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Theia Clinical Research, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Midway Specialty Care Center, West Palm Beach, Florida
  - Cleveland Clinic, Weston, Florida
  - Flourish Research, Winter Park, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - Medster Research, Valdosta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Infectious Disease Consultants Clinical Research, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Northwell Health, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai-National Jewish Respiratory Institute, New York, New York
  - Columbia University, New York, New York
  - NYC Health and Hospitals-Elmhurst, Queens, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Temple Lung Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Low Country Infectious Diseases, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - The University of Texas Health Science Center, Tyler, Texas
  - UVA Health Infectious Diseases Clinic, Charlottesville, Virginia
- Australia (9):
  - Macquarie University Clinical Trials Unit, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Monash University Centre for Inflammatory Diseases, Cranbourne, Victoria
  - Alfred Health, Melbourne, Victoria
  - Royal Perth Hospital Respiratory Clinic, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Concord Repatriation General Hospital, Concord
- Japan (25):
  - Aso Iizuka Hospital, Fukuoka
  - National Hospital Organization Fukuokahigashi Medical Center, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Fukuoka University Chikushi Hospital, Fukuoka
  - National Hospital Organization Omuta National Hospital, Fukuoka
  - National Hospital Organization Shibukawa Medical Center, Gunma
  - Himeji Medical Center, Hyōgo
  - Ibarakihigashi National Hospital, Ibaraki
  - Kameda Clinic, Kamogawa-shi
  - SHOWA University Fujigaoka Hospital, Kanagawa
  - Minami Kyoto Hospital, Kyoto
  - Matsusaka Municipal Hospital, Matsusaka
  - Sendai Kousei Hospital, Miyagi
  - Nishiniigata Chuo Hospital, Niigata
  - National Hospital Organization - Osaka Toneyama Medical Center, Osaka
  - Saitama Prefectural Cardiovascular and Respiratory Center, Saitama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Keio University Hospital, Shinjuku-ku
  - National Hospital Organization Tenryu Hospital, Shizuoka
  - Mutual Aid Associations Toranomon Hospital, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Japanese Red Cross Musashino Hospital, Tokyo
  - Japan Anti-Tuberculosis Association Fukujuji Hospital, Tokyo
  - SHOWA University Northern Yokohama Hospital, Yokohama
- South Korea (6):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
- Taiwan (5):
  - National Taiwan University Hospital, Hsinchu
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei